CLINICAL TRIAL: NCT03259776
Title: Experiences of Visitors to a Regional Major Trauma Intensive Care Unit
Acronym: VISIT_ICU
Status: Completed | Type: Observational
Sponsor: Kingston University (Other)
Responsible Party: Principal Investigator, Stefan Tino Kulnik, Postdoctoral Researcher, Kingston University
Other Study IDs: 233327
Record Dates: First submitted 2017-08-17; First posted 2017-08-24 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Major Trauma
Keywords: Intensive Care; Patient- and Family-Centred Care; Patient and Public Involvement; South West London Major Trauma Network; Service Improvement; Survey Questionnaire; Visitor Experiences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Visitors: Qualitative interviews and questionnaire survey
  Interventions: Other: Qualitative interviews and questionnaire survey

INTERVENTIONS:
Other: Qualitative interviews and questionnaire survey — Qualitative interviews and questionnaire survey

SUMMARY:
Since 2011, people who have had a serious accident in England are no longer looked after at the hospital nearest to them. Instead, they are cared for at a specialist hospital called the regional major trauma centre. This is so that they can get the best possible care from specialist professionals.

St George's is the regional major trauma centre for the 2.6 million people living in South West London and Surrey County. This area stretches about 40 miles across.

About one fifth of major trauma patients who come to St George's live more than one hour's journey away. Their visitors often travel a similar distance or even further. Family members and friends play an important part during the patient's stay. It is important to support visitors.

The aim of this study is to describe the experiences of visitors whose family member or friend has been admitted to the major trauma intensive care unit at St George's. In particular, the aim is to describe the experiences of visitors who travel from far.

First, ten visitors will be interviewed to find out more about their experiences. From these data, a survey questionnaire will then be developed and approximately 150 visitors who have been to St George's in recent months will be surveyed. This will give in-depth insights to understanding peoples' experiences of visiting at St George's, and what people thought was going well and things that could be better. The study will end with a service improvement workshop with representatives from the team at St George's and visitors. Study findings will be discussed and decisions on what should be improved will be made.

This study is being funded by St George's Hospital Charity. The study runs from August 2017 to October 2018.

ELIGIBILITY:
Inclusion Criteria:

* Visitors (i.e. designated next of kin and/or other family member or friend with a close relationship and significant involvement in the patient's circumstances and care) of a patient who has been admitted to intensive care at St George's University Hospitals NHS Foundation Trust under the major trauma care pathway
* Ordinary residence further away than one hour's drive from St George's Hospital (estimated driving time in mid-week mid-morning traffic according to Google Maps, equating to a distance of approximately 30 miles)
* Adults (18 years and over)
* Written informed consent (for semi-structured qualitative interviews)

Exclusion Criteria:

* Ordinary residence within one hour's drive from St George's Hospital (estimated driving time in mid-week mid-morning traffic according to Google Maps, equating to a distance of within approximately 30 miles)
* Limited English (for semi-structured qualitative interviews)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visitors (i.e. designated next of kin and/or other family member or friend with a close relationship and significant involvement in the patient's circumstances and care) of a patient who has been admitted to ICUs at St George's University Hospitals NHS Foundation Trust under the major trauma care pathway
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Visitors' experiences | 15 months
  This study uses mixed-methods in a two-staged approach, to provide both depth and breadth in capturing data on visitors' experiences.
  In the first stage, a series of semi-structured qualitative interviews will capture in-depth data on visitors' experiences. Participants will be asked questions such as "Can you talk a bit about visiting your relative/friend here at St George's" and "How has your daily life been since you started visiting here at St George's". These in-depth qualitative data will inform the content and structure for a bespoke visitor experience questionnaire, which will be newly developed as part of the study and copyrighted.
  In the second stage, the newly developed, bespoke visitor experience questionnaire will be used to survey a larger number of visitors, gathering both quantitative and qualitative data to describe the experiences of visitors, areas of good practice and needs and opportunities for service improvement at the study site.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan T Kulnik, PhD, Principal Investigator — Kingston University
Locations (1):
- St George's University Hosptials NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No